CLINICAL TRIAL: NCT05787639
Title: Neoadjuvant Radiation and Evorpacept (ALX148) in Combination With Pembrolizumab In Patients With Previously Untreated Locally Advanced, Resectable, HPVOPC (Human Papilloma Virus Oropharynx Cancer)
Brief Title: Neoadjuvant Immunoradiotherapy With Evorpacept and Pembrolizumab in HPVOPC (Human Papilloma Virus Oropharynx Cancer)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Joseph Califano, Professor, Department of Otolaryngology-Head and Neck Surgery, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 806684
Record Dates: First submitted 2023-02-28; First posted 2023-03-28 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-05

CONDITIONS: Oropharynx Cancer
MeSH Terms: conditions — Oropharyngeal Neoplasms | interventions — ALX148

STUDY DESIGN:
Intervention Model Description: A phase II clinical trial for AJCC (American Joint Committee on Cancer) VIII Stage I T1-2N1M0 HPVOPC, including patients amenable to surgical resection, excluding patients with solitary lymph nodes less than 3 cm who are amenable to surgical therapy alone. Stereotactic radiation therapy (SBRT (8GyX3)) will be delivered to gross tumor volume (GTV) +3mm, followed by Pembrolizumab 200 mg IV and Evorpacept 45 mg/kg IV every three weeks x 2 cycles followed by surgical resection of primary tumor and neck dissection. The primary endpoint is pathologic response compared to historical standard of care rates of locoregional control, and secondary endpoints are clinical response, survival, and safety and toxicity.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental): Stereotactic radiation therapy (SBRT (8GyX3)) will be delivered to gross tumor volume (GTV) +3mm, followed by Pembrolizumab 200 mg IV and Evorpacept 45 mg/kg IV every three weeks x 2 cycles followed by surgical resection of primary tumor and neck dissection.
  Interventions: Drug: Evorpacept

INTERVENTIONS:
Drug: Evorpacept — After stereotactic radiation to primary tumor and neck on week 1 of study, Evorpacept 45 mg/kg is administered by IV infusion every three weeks starting on Week 2, Day 1 of study for a total two 21-day cycles (6 weeks)
  Other Names: ALX 148

SUMMARY:
The majority of head and neck cancer patients do not respond to immunotherapies, and clinical responses are often not durable. However, targeting tumors with stereotactic radiation in combination with immunotherapy while sparing draining lymphatics enhances anticancer immunity, resulting in dramatic response in HPV (Human Papilloma Virus) virus related cancers of the throat. This trial will leverage targeted tumor radiation and immunotherapy in advance of standard surgical therapy to improve the response of HPV (Human Papilloma Virus) throat cancer to radiation and immunotherapy.

DETAILED DESCRIPTION:
This is a prospective, multi-center, open-label, one-arm, two-stage, Phase II study to evaluate the efficacy of neoadjuvant immunoradiotherapy (NIRT) in patients with stage I HPVOPC (Human Papilloma Virus Oropharynx Cancer) amenable to surgical resection, including AJCC (American Joint Committee on Cancer) VIII T1-2N1M0 HPVOPC (Human Papilloma Virus Oropharynx Cancer) and excluding patients with solitary lymph nodes less than 3 cm. A Simon's two-stage optimal design is used for this study. We will test the hypothesis that neoadjuvant stereotactic tumor targeting radiation along with CD47 inhibition (evorpacept) and PD-1 inhibition (pembrolizumab) provides pathologic response compared to current standard of care rates of locoregional control.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of Stage I T1-2N1M0 HPVOPC (Human Papilloma Virus Oropharynx Cancer)
* Amenable to surgical resection
* Are able to safely receive neoadjuvant radiation and Evorpacept/Pembrolizumab

Exclusion Criteria:

• Patients with solitary lymph nodes less than 3 cm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2024-02-20 (Actual); Primary Completion 2026-08-20 (Estimated); Study Completion 2028-05-30 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response | week 7-10
  Pathologic response is determined when surgery is performed at week 7-10 of study
Major pathologic response | week 7-10
  Major pathologic response is defined as <10% viable tumor cells in the resection specimen) after surgical resection

SECONDARY OUTCOMES:
clinical response | week 7
  clinical response will be determined by clinical and radiographic criteria by comparison of pretreatment and post-treatment assessment prior to surgery
clinical to pathologic down-staging | week 7-10
  clinical to pathologic down-staging will be assessed by comparing pretreatment AJCC (American Joint Committee on Cancer) VIII stage to pathologic stage determined by surgical pathology results. And decrease in overall Stage or decrease in T or N category will be defined as down staging.
overall survival | 3 years
  survival will be determined based on intent to treat analysis at conclusion of study after 3 years
disease free survival | 3 years
  subjects will be assessed for presence of disease after completion of treatment and up to three years
Safety and toxicity | 11 months to three years
  Safety and toxicity will be assessed by CTCAE for overall toxicity and safety and Clavien-Dindo for toxicity related to surgery.
Patient-reported quality of life and functional outcomes (score 0-100 with 100 being best possible score) | post treatment at 7, 11 weeks and at 3 and 12 months
  The University of Washington-Quality of Life (UW-QOL) to assess standard penetration-aspiration score (PAS) will be used to assess patient and observer-reported quality of life and functional outcomes.
Patient-reported quality of life and functional outcomes (score 20-100 with 100 being best possible score) | post treatment at 7, 11 weeks and at 3 and 12 months
  MD Anderson Dysphagia Inventory (MDADI) to assess standard penetration-aspiration score (PAS) will be used to assess patient and observer-reported quality of life and functional outcomes.
Observer-reported quality of life and functional outcomes | post treatment at 7, 11 weeks and at 3 and 12 months
  Video Fluoroscopic Swallow Study (VFSS) to assess standard penetration-aspiration score (PAS) will be used to assess patient and observer-reported quality of life and functional outcomes.
Immune Correlates (T-cell infiltration) | 7-11 weeks
  Patients will undergo assessment of T-cell infiltration into primary tumors expressed as % staining in primary tumor sections on immunohistochemical staining.
Immune Correlates (shared tumor and sentinel node T-cell clones) | 7-11 weeks
  Patients will undergo assessment of frequency of shared tumor and sentinel node T-cell clones as defined by absolute number of shared clones,
Immune Correlates (B-cell germinal centers) | 7-11 weeks
  Patients will undergo assessment of number of B-cell germinal centers in draining sentinel lymph nodes compared to non-sentinel nodes as defined by average number of B-cell germinal centers per high powered field with random sampling of at least 10 high powered fields on microscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Jospeh A Califano, MD, Principal Investigator — University of California, San Diego
Locations (3):
- United States (3):
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Providence Health & Services, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mombelli A. [Periodontal diagnosis. The role of microbiology]. Schweiz Monatsschr Zahnmed. 1994;104(1):48-57. No abstract available. French, German. PMID 8108690
- See also: This publication presents phase I data supporting a neoadjuvant immunoradiotherapy approach for HPVOPC (Human Papilloma Virus Oropharynx Cancer), demonstrating 90% pathologic complete response. — https://pubmed.ncbi.nlm.nih.gov/33963014/